CLINICAL TRIAL: NCT03161587
Title: Patient Characteristics and Treatment Modalities in COPD Patients Assessed by GOLD2016 : a Cross-Sectional Study in China
Brief Title: Patient Characteristics and Treatment Modalities in COPD Patients in China
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207136
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: FEV1; COPD; CAT; treatment modality; FVC; GOLD 2016; mMRC
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with COPD: Subjects with diagnosis of COPD at least one year, visiting outpatient clinics in tertiary hospitals in China and in stable state at enrolment.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a complex disease characterized by multiple clinical manifestations as well as co-morbidities. While COPD subjects have traditionally been classified based solely on airflow limitation (forced expiratory volume in one second [FEV1]), a new classification system was introduced in the year of 2011 by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) that recommended subjects with COPD should be classified based on a combination of airflow limitation, disease impact (determined by symptom burden and activity limitation) and history of exacerbation. This approach results in the classification of subjects in four groups: A (low risk, less symptoms), B (low risk, more symptoms), C (high risk, less symptoms), and D (high risk, more symptoms). This classification system was further refined in year 2013, specifically around the history of exacerbation definition, where having ≥1 exacerbation leading to hospital admission in preceding year was added as a criteria for classification into the "high risk" C or D groups. Further, in the year 2016, there was a refinement of the disease impact criteria that suggest the use of the COPD Assessment Test (CAT) score (over the Modified British Medical Research Council Dyspnea Scale [mMRC] score) as the preferred tool to determine classification as "more symptoms" or "less symptoms". This study aims to understand subject characteristics and current treatment modalities in different groups classified by GOLD 2016 comprehensive classification system and to understand if current treatment choice is concordant with the GOLD recommendations in real life clinical practice in China tertiary hospitals. It will provide a useful point-in-time description of COPD subject characteristics and current treatment modalities in real life clinical practice in China.

ELIGIBILITY:
Inclusion criteria

* Aged 40 years and older
* A clinical diagnosis of COPD for at least one year: dyspnea, chronic cough or sputum production, and a history of exposure to risk factors for the disease and lung function test FEV1/ FVC <0.7(post bronchodilator)
* Out-patient
* Able to read, comprehend, and record information in Chinese
* A signed and dated written informed consent must be obtained from the subject prior to study participation Exclusion criteria
* Current exacerbation or an exacerbation within the preceding one month
* Other unstable diseases which could influence CAT and lung function results (judged by physicians)
* A medical diagnosis of active tuberculosis, cystic fibrosis, any other pulmonary condition, lung cancer, or hypereosinophilic syndromes (HES)
* Currently participating in another COPD clinical study which provides the subject investigational medication and/or disease management

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of COPD subjects who are being managed for their disease at outpatient clinics in tertiary hospitals. Subjects diagnosed with COPD for at least one year and in the stable state at enrolment with no exacerbation events in the preceding month are included.
Sampling Method: Probability Sample
Enrollment: 848 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects classified into each of the GOLD 2016 comprehensive classification system groups | Day 1
  Subjects will be classified into groups A-D according to GOLD 2016 comprehensive classification system. Symptoms will be assessed with the CAT scale to determine if the subject belongs to the boxes of side-Less Symptoms (CAT <10) or side-More Symptoms (CAT ≥10).
  Risk of exacerbations will be assessed to determine if the subject belongs to the lower part of the box-Low Risk or the upper part of the box-High Risk.
  Spirometry will be used to determine the GOLD grade of airflow limitation (GOLD 1 and GOLD 2 categories indicate Low Risk, while GOLD 3 and GOLD 4 indicate High Risk).
To determine the demographic characteristics for each GOLD 2016 group | Day 1
  Subject's height, weight and waistline will be measured. Body Mass Index will be calculated by height and weight, and smoking status will be reported and recorded.
To determine co-morbid diseases | Day 1
  Cardiovascular diseases (ischemic heart disease, heart failure, atrial fibrillation, hypertension), diabetes, hyperlipidemia, anxiety, depression, gastroesophageal reflux disease (GERD), obstructive sleep apnea syndrome (OSAS), bronchiectasis, allergic airway disease be reported and recorded.
To assess the disease severity by CAT score | Day 1
  Symptom assessment will be done based on CAT score. The CAT is a validated, short and simple subject completed questionnaire which has been developed for use in routine clinical practice to measure the health status of subjects with COPD. Subjects are scored on eight items (cough, phlegm, chest tightness, breathlessness, activity limitation, confidence, sleep and energy) on a scale of 0-5 depending on their impact. The sum of scores for each item gives the subject's impact score ranging from 0 (no impact) to 40 (worst possible impact). Subjects will be stratified as score < 10 and ≥10.
To assess the disease severity by lung function | Day 1
  Subjects will undergo a lung function test (FEV1 and Forced Vital Capacity [FVC]) during the study visit if they do not have record of a lung function test report in last 6 months.
No of subjects with exacerbation history and hospitalization for exacerbation in preceding year | Day 1
  An exacerbation of COPD is an acute event characterized by a worsening of the subject's respiratory symptoms that is beyond normal day-to-day variations and leads to a change in medication. Subject's exacerbation history in the preceding year will be measured and recorded on the subject note

SECONDARY OUTCOMES:
Number of subjects treated in concordance with first and alternative choice treatments recommended for each GOLD 2016 grade based on current maintenance treatment | Day 1
  GOLD 2016 A-D group's current maintenance treatment will be regarded as concordant with "Recommended First Choice" if subject's current maintenance treatment is one of "recommended first choice" for his/her group. By the same rule, a subject's current maintenance treatment will be regarded as concordant with "alternative choice" if his/her current maintenance is one of "alternative choice" for his/her group.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- China (8):
  - GSK Investigational Site, Xiamen, Fujian
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Hohhot, Inner Mongolia
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Zhengzhou